CLINICAL TRIAL: NCT05463380
Title: Hospitalised COVID-19 Patients Cohort Study in the EuCARE Project
Acronym: EuCARE-HOSP
Status: Recruiting | Type: Observational
Sponsor: Euresist Network GEIE (Other)
Collaborators: Karolinska Institutet (Other); Centro Hospitalar Lisboa Ocidental (Other Government); Heinrich-Heine University, Duesseldorf (Other); ASST Santi Paolo e Carlo (Other); Imperial College London (Other); Vilnius University Hospital Santaros Klinikos (Other); University of Rome Tor Vergata (Other); Bach Mai Hospital (Other); Kenya Medical Research Institute (Other); Hospital Regional de Alta Especialidad "Dr. Juan Graham Casasus" (Other); University Hospitals Dorset NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: EuCARE-HOSPITALISED study
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — biological material from COVID-19 in-patients in a diverse setting of 12 hospitals/clinics in 11 countries and 4 continents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized COVID 19 patients: Hospitalized adult (>18 years) patients including patients in the emergency ward Positive for SARS-CoV-2 by PCR any time from 14 days before admission date until hospital discharge. Both first and recurrent episodes of COVID-19 will be included.
  Having a signed informed consent when required by ethical approval
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — The patient will be treated following the satndard of care in the participating units

SUMMARY:
The WP3 hospitalized cohort in EuCARE is an observational multicentre study including collection of retrospective (historical) and prospective data from hospitalized COVID-19 patients followed at 12 clinics from 11 countries from 4 continents. In a subset of patients, peripheral blood, viral isolates and/or viral sequences are collected for analysis in WP2 with regards to neutralising antibodies, cellular immunity and SARS-CoV-2 diagnostics. Data and results from analysis of biological material will be analysed by biostatistical methods and with artificial intelligence in WP5. This analysis will focus on the impact on clinical outcome of viral variants / viral sequences as well as the vaccines used and the vaccination schedules.

DETAILED DESCRIPTION:
Background: Since the start of the COVID-19 pandemic, novel SARS-CoV-2 variants of concern have emerged, some of which have become largely dominant including the B.1.1.7 (alpha), the B.1.617 (delta) and more recently the B.1.1.529 (omicron). The clinical implications of the different variants in unvaccinated and vaccinated persons are still not adequately characterized. The detailed understanding of the interplay between the variants, vaccine immune responses and disease severity is still scarce.

Study objectives:

Overall objectives are:

* to collect data and/or biological material from COVID-19 in-patients in a diverse setting of 12 clinics in 11 countries and 4 continents
* to analyse the clinical course of COVID-19 in in-patients in relation to the viral characteristics
* to analyse the clinical course of COVID-19 in in-patients in relation to vaccines used and vaccination schedules
* to deliver recommendations for optimized clinical management and treatment with special consideration to viral characteristics and to used vaccines

Specific objectives are:

* To describe the patterns of clinical symptoms, therapeutic interventions and clinical outcome in patients hospitalized from 12 hospitals/clinics, in 11 countries and 4 continents.
* To assess the impact of viral variants / viral sequences on the clinical outcome measured as all-cause in-hospital mortality, non-invasive mechanical ventilation/high-flow nasal oxygen, mechanical ventilation, admission to intensive care unit, length of time in intensive care and overall length of hospitalization.
* To assess the impact of different vaccines and vaccination schedules on the clinical outcome measured as all-cause in-hospital mortality, non-invasive mechanical ventilation/high-flow nasal oxygen, mechanical ventilation, admission to intensive care unit, length of time in intensive care and overall length of hospitalization.
* To assess the impact of viral variants / sequences in response to treatment interventions and the associated clinical outcome
* To assess the impact of different vaccines and vaccination schedules in response to treatment interventions and the associated clinical outcome
* To provide WP2 in EuCARE with biological material for further studies on viral characteristics and associated immune responses
* To provide WP5 in EuCARE with data for further studies using artificial intelligence

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult (>18 years) patients including patients in the emergency ward
* Positive for SARS-CoV-2 by PCR any time from 14 days before admission date until hospital discharge. Both first and recurrent episodes of COVID-19 will be included.
* Having a signed informed consent when required by ethical approval

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult (>18 years) patients including patients in the emergency ward Positive for SARS-CoV-2 by PCR any time from 14 days before admission date until hospital discharge. Both first and recurrent episodes of COVID-19 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
Severity of SARS-CoV-2 infection | through study completion, an average of 4 year
  This is currently being discussed, which classification system should be used. This will be harmonized to recommendations by the WHO/ISARIC or other source.
In-hospital mortality | through study completion, an average of 4 year
  YYYY-MM-DD or NA if discharged alive
ICU Admissions and Discharges | through study completion, an average of 4 year
  YYYY-MM-DD or NA if not ICU-admitted
Rate of Invasive and Non invasive mechanical ventilation | through study completion, an average of 4 year
  Yes/No/Unknown - If yes, duration of mechanical ventilation

SECONDARY OUTCOMES:
Frequency and type of Renal replacement therapies (RRT, dialysis) | through study completion, an average of 4 year
  Yes/No/Unknown
Frequency of Blood transfusions | through study completion, an average of 4 year
  Yes/No/Unknown
Frequency of ECMO Frequency of ECMO | through study completion, an average of 4 year
  Yes/No/Unknown

CONTACTS AND LOCATIONS:
Overall Officials: ANDERS Sönnerborg, Prof, Study Chair — Karolinska Institutet
Locations (10):
- Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany
- Italy (2):
  - ASST Santi Paolo e Carlo, Milan, Lombardy
  - University of Rome Tor Vergata, Rome
- Kenya Medical Research Institute (KEMRI), Nairobi, Kenya
- Vilnius universiteto ligoninė Santaros klinikos, Vilnius, Lithuania
- Regional Hospital Dr. Juan Graham Casasús, Villahermosa, Villahermosa, Mexico
- Centro Hospitalar Lisboa Ocidental, Lisbon, Portugal
- Karolinska Institutet, Stockholm, Sweden
- Poole University Hospitals, Dorset, Poole, United Kingdom
- Bach Mai Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The study is part of a project funded by the European Commission and the project agreement with the Commission affirms that the data and the results will be publi
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: AFTER THE STUDY END NO TIME LIMIT WAS FIXED
Access Criteria: REQUEST TO THE STUDY COORDINATOR OR TO THE PROJECT PARTNERS
URL: https://eucareresearch.eu/

REFERENCES:
- [Derived] Hedberg P, Varisco B, Bai F, Sonnerborg A, Naucler P, Pfeifer N, Cozzi-Lepri A, Ceccherini-Silberstein F, Naumovas D, Drobniewski F, Jensen BO, Toscano C, Parczewski M, Quintanares GHR, Mwau M, Pinto JA, Incardona F, Mommo C, Marchetti G. EuCARE-hospitalised study protocol: a cohort study of patients hospitalised with COVID-19 in the EuCARE project. BMC Infect Dis. 2023 Oct 16;23(1):690. doi: 10.1186/s12879-023-08658-2. PMID 37845624